CLINICAL TRIAL: NCT00000350
Title: Effects of Stimulant Dependence on Human Striatal Dopamine System
Brief Title: Effects of Stimulant Dependence on Human Striatal Dopamine System - 15
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: NIDA-3-0010-15; Y01-3-0010-15
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 1999-03

CONDITIONS: Amphetamine-Related Disorders; Tobacco Use Disorder
Keywords: amphetamine dependence
MeSH Terms: conditions — Amphetamine-Related Disorders; Tobacco Use Disorder

INTERVENTIONS:
Procedure: radioactive substance

SUMMARY:
The purpose of this study is to determine whether DAT availability, assessed by WIN binding, in the striatum is altered in cocaine or methamphetamine dependence. To determine whether DA synthesis capacity, assessed by FDOPA uptake, in the striatum is altered in Coc or Meth dependence. To determine whether the PET tracers, WIN or FDOPA, will differentiate Meth induced alterations from those induced by Coc use. To determine whether the PET characterization of striatal alterations observed at 3-5 days since last drug use persists at least 3 months after last drug use.

DETAILED DESCRIPTION:
4-5 Day inpatient study. Participant will have scanned pictures (MRI & PET scans) taken of their brain after being injected with a small amount of WIN, a radioactive substance. Participants give daily urine samples and fill out health related questionnaires. It is important to determine whether the alterations characterized within one week of last drug use persist over a longer time period. Based on results of the studies from aims 1 & 2, we will decide which of the 2 probes, WIN or FDOPA-PET is the more sensitive index of stimulant-dependency-induced changes.

ELIGIBILITY:
Inclusion Criteria:

M/F, ages 21-50. Meet DSM-IV criteria for methamphetamine and nicotine dependence. Agree to conditions of the study and sign informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy. History of seizures. Pregnant and/or nursing women. Dependence on ETOH or benzodiazepines or other sedative/hypnotics. Acute hepatitis. Other medical conditions that deem participation to be unsafe.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1999-03

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States